CLINICAL TRIAL: NCT04945291
Title: Evaluation of a Food Estimation Method Using the Hands and a Mobile App for Self-monitoring of Calories and Weight Loss: a Randomized Controlled Trial
Brief Title: Calories Counting Using an App for Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Jumana Antoun, Associate Professor of Family Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBS-2021-0041
Record Dates: First submitted 2021-06-17; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: three- armed randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The participants will know the application they are using; the outcome assessor will be blinded to the user app when they fill the questionnaire and take the height and weight measurements
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- research built JA Method mobile application + Counting method using the hands (Experimental): The participant will watch a video that explains a new counting method using the hands and use the research built mobile application to log and track the calories
  Interventions: Behavioral: New way of counting calories using the hands; Behavioral: Mobile applications
- FitnessPal mobile application (or Arabic alternative) + Counting method using the hands (Active Comparator): the participants will watch a video that explains a new counting method using the hands and they will be asked to use a commercial mobile app to log and track the calories
  Interventions: Behavioral: New way of counting calories using the hands; Behavioral: Mobile applications
- Fitness Pal Mobile Application (or Arabi alternative) (Active Comparator): The participants will watch a generic video about the mobile app and they will be asked to use a commercial mobile app to log and track the calories
  Interventions: Behavioral: Mobile applications

INTERVENTIONS:
Behavioral: New way of counting calories using the hands — The participants will learn how to estimate the portions and calories content of food using their hands as a measurement tool;
  Arms: FitnessPal mobile application (or Arabic alternative) + Counting method using the hands; research built JA Method mobile application + Counting method using the hands
Behavioral: Mobile applications — the participant will use a mobile application to log their calories

SUMMARY:
This research aims to measure anew way of calories counting using a mobile app on weight loss and adherence to the mobile app. The participants should be adults who is overweight or obese and should have a smartphone with access to the internet. The participants will fill a baseline survey, take the height and weight measurements, watch a video about the use of the calories counting and app. A follow up visit will be in 4 weeks to take the height and weight measurements and fill a questionnaire. There is an option for the participants to continue with the research for additional 11 months with visit at 3, 6 and 12 months.

DETAILED DESCRIPTION:
Obesity has been recognized as a disease by the American Medical Association in 2013. It has been alarmingly on the rise over the past two decades, especially in the MENA region. In Lebanon, 53.5% of the population is overweight and 18.16% obese. Self-monitoring, as part of behavioral interventions, is beneficial for weight loss, especially in the context of mobile application interventions. However, estimation of the food portions for proper food logging remains a challenge despite the use of databases, scales and household utensils.

Objective: To measure the efficacy of a novel 12-month self-monitoring program for weight loss and long-term adherence to the use of the application. The program entails estimation of food consumption using the hand and a mobile application (developed by the research team) that relies on evidence-based behavioral interventions.

Design: Randomized controlled trial Setting: American University of Beirut Medical Center Participants: Adults who are overweight or obese will be recruited from AUB/AUBMC staff and students and the community. Participants should be 18 years old and above and should have a smartphone with access to the internet.

Interventions: This research will be a three-armed randomized controlled trial. The first phase (I) will test three different methods of calorie counting each allocated to an arm of our trial at 4 weeks and the second phase (II) will test the long term efficacy of our method and its sustainability. One arm specific for the control group will be using a commercial mobile application called Fitness Pal (or رشاقة for Arabic preference) alone; another arm will be using the commercial mobile application Fitness Pal (or رشاقة for Arabic preference) along with the food estimation method using hands, and the third arm will be using the developed mobile application of the study along with the food estimation method using hands. Phase I constitutes a baseline and 4-weeks-visit where we will seek the participants' feedback concerning the mobile application and the hand counting method. Phase II: participants who are motivated to continue using the mobile applications and self-monitoring will be followed up to a period of one year.

Follow up visits will take place at 3 months, 6 months, and 12 months following the start of trial to assess for any change in participant's weight and adherence to the use of the mobile application and counting method.

Main Outcome Measures: The primary outcome of phase I will be the satisfaction with the counting method and mobile app mobile application rating and satisfaction with the various application features. The primary outcome of phase II will be the difference in the percentage of participants who achieved weight loss of 5% of their baseline weight among the three groups at 3 months, 6 months, and weight loss of 10% of their baseline weight at 12 months post-intervention.

Secondary outcomes include (1) a decrease in weight in Kg from baseline at 1,3,6 and 12 months; (2) a decrease in waist circumference in cm from baseline at 1, 3, 6, and 12 months, (3) frequency of logging in days, (4) adherence to the use of the application. In addition, demographics characteristics, self-regulation and internal motivation of the participants will be explored whether they affect any of the primary and secondary outcomes

ELIGIBILITY:
Inclusion Criteria:

* Should have a smartphone with access to the internet
* BMI more than 25 (overweight or obese)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieved weight loss of 5% of the baseline weight | 3 months

SECONDARY OUTCOMES:
UMARs satisfaction scores | 1 month
  Satisfaction with the mobile application features
Percentage of participants who achieved weight loss of 5% of their baseline weight | 6 months
Percentage of participants who achieved weight loss of 10% of their baseline weight | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jumana Antoun, Hamra, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No